CLINICAL TRIAL: NCT07103785
Title: The Effectiveness of a Mobile Game Intervention in Modifying Attentional Bias Toward Alcohol Cues: A Randomized Controlled Trial
Brief Title: The Effectiveness of a Mobile Game Intervention in Alcohol Use Disorder
Acronym: Gamification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zehra Su Topbaş, research assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2011-KAEK/80
Record Dates: First submitted 2025-07-24; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder
Keywords: attentional bias; modification; mobile app; gamification
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 30 patients who met the inclusion and exclusion criteria.
  Interventions: Drug: Akamprosat or Naltrekson or combined medical treatment (Akamprosat and Naltrekson)
- Mobile game group (Experimental): 30 patients who met the inclusion and exclusion criteria.
  Interventions: Other: Mobile game app; Drug: Akamprosat or Naltrekson or combined medical treatment (Akamprosat and Naltrekson)

INTERVENTIONS:
Other: Mobile game app — The mobile game designed to modify attentional bias toward alcohol-related cues was developed by integrating game elements into a modified version of the dot-probe task. This gamified intervention was installed on the smartphones of participants assigned to the experimental group, and each participant was provided with a unique username and password for access. Participants were instructed to engage with the mobile game every other day over one month.
  Arms: Mobile game group
Drug: Akamprosat or Naltrekson or combined medical treatment (Akamprosat and Naltrekson) — Medicines prescribed by a doctor for the treatment of Alcohol Use Disorder (Akamprosat or Naltrekson or combined medical treatment (Akamprosat and Naltrekson))

SUMMARY:
The aim of this study was to evaluate the effectiveness of a mobile game application targeting attentional bias modification for alcohol stimuli in patients with Alcohol Use Disorder. Attentional bias is the tendency for individuals to pay more attention to some environmental stimuli than others. Previous evidence suggests that attentional bias for alcohol stimuli is associated with severity of drinking and craving. The research questions are as follows;

* Does the developed mobile game application reduce the attentional bias related to alcohol?
* Does the developed mobile game application reduce alcohol craving severity?
* Does the developed mobile game application reduce the severity of alcohol drinking? The researchers will evaluate the effectiveness of the mobile game, which aims to reduce attentional bias to alcohol stimuli, as standard treatment for Alcohol Use Disorder (medical treatment) versus standard treatment + mobile game application group.

Participants,

* Comply with the medical treatment prescribed by the doctor
* Use the mobile gaming app every other day for one month
* Come back in a month for an evaluation
* Be available for a telephone interview three months after the first interview

DETAILED DESCRIPTION:
Alcohol Use Disorder (AUD) is a significant public health problem that has far-reaching consequences for the well-being of individuals, families, and society. Recent studies have demonstrated that attentional bias for alcohol-related stimuli is associated with several variables, including alcohol craving, alcohol consumption behavior, and relapse following treatment. Therefore, interventions aimed at modifying attentional bias for alcohol cues have been a subject of scholarly interest.

The literature shows that, in addition to psychotherapeutic strategies, computerized versions of conventional attentional bias assessment instruments-referred to as Attentional Bias Modification (ABM)-have been utilized to decrease alcohol-related attentional bias. Some research indicates that ABM training produces results similar to psychotherapeutic treatments. ABM has the benefits of fewer interaction demands, time, and geographical limitations.

Gamified ABM methods have displayed encouraging impacts in decreasing craving, substance use, and relapse in different types of addiction. Nevertheless, research assessing gamified ABM treatments in people specifically diagnosed with AUD is still limited. Due to this shortage, an investigation of the effectiveness of gamified ABM treatments for AUD is deemed both timely and essential. Notably, most current ABM games for AUD have been created for desktop and laptop computers. Considering the extensive availability of mobile devices, providing such treatments through mobile devices will likely boost reach and user acceptance.

To meet these requirements, the current study created a gamified mobile ABM treatment to decrease attentional bias for alcohol cues in patients diagnosed with AUD. In the first phase, qualitative content analysis was gathered, and expert and patient feedback on the game was analyzed. The game was adjusted, and its final version was prepared according to this feedback.

The game's efficacy was tested in a tertiary care hospital in a northwestern province of Türkiye. Sixty subjects were enrolled-30 in the intervention group and 30 in the control group. All the subjects were given standard medical therapy as prescribed by a physician. Besides, the intervention group was also asked to use the mobile game developed for altering alcohol-related attentional bias. They were told to play the game every other day for a month.

The participants filled out the Penn Alcohol Craving Scale (PACS), the Alcohol Use Disorders Identification Test (AUDIT), and the Dot-Probe Task as pre- and post-tests. Three months following the post-test, follow-up data were gathered through phone interviews. Statistical analysis through chi-square tests, independent samples t-tests, and linear mixed models will be used to assess intervention efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Ability to speak and understand Turkish
* Literacy (reading and writing)
* Ability to use a smartphone
* Having received a formal diagnosis of Alcohol Use Disorder (AUD)
* Receiving outpatient treatment and follow-up care for AUD
* Scoring 8 or higher on the Alcohol Use Disorders Identification Test (AUDIT)

Exclusion Criteria:

* Currently experiencing an active psychotic episode
* Currently in a manic or hypomanic episode
* Having a neurodevelopmental or neurocognitive disorder
* Exhibiting symptoms of delirium
* Being under the influence of alcohol or other substances to a degree that negatively affects cognitive functioning
* Having participated as a qualitative data contributor in the initial phase of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Dot-Probe Task | Average 30 days: measurement before intervention (Time 1), 4 weeks after intervention, immediately after intervention measurement (Time 2)
  The Dot-Probe Task was used to assess attentional bias toward alcohol cues. The procedure was built using E-Prime 3.0 and conducted via laptop. Each trial began with a fixation cross (1000 ms), followed by alcohol-neutral image pairs for another 500 ms, displayed on opposite sides of the screen. Ninety-two culturally relevant beverage images (46 alcohol, 46 non-alcohol) were used, including beer, wine, rakı, whiskey, water, soda, cola, and iced coffee. The experiment consisted of three blocks of 46 trials. Participants were instructed to identify the location of a probe, appearing where one image had been, by pressing the left or right arrow key as quickly as possible. A four-trial practice block preceded the task. Reaction time differences between probes replacing alcohol vs. neutral cues were used to calculate attentional bias scores. Higher bias scores indicated increased attention toward alcohol-related stimuli.

SECONDARY OUTCOMES:
The Penn Alcohol Craving Scale (PACS) | Average 30 days: pre-intervention measurement (Time 1), 4 weeks intervention, immediately after the intervention measurement (Time 2), Three months after Time 2 (Time 3)
  The Penn Alcohol Craving Scale (PACS) is a self-report instrument to assess the intensity of alcohol craving during the past week. It evaluates five dimensions of craving: frequency, intensity, duration, resistance, and overall craving. The scale consists of five items under a single subdimension. Each item is scored on a scale from 0 to 6, yielding a maximum total score of 30. Higher scores indicate greater levels of alcohol craving.
The Alcohol Use Disorders Identification Test (AUDIT) | Average 30 days: pre-intervention measurement (Time 1), 4 weeks intervention, immediately after the intervention measurement (Time 2), Three months after Time 2 (Time 3)
  The Alcohol Use Disorders Identification Test (AUDIT) is a 10-item questionnaire designed to gather information on alcohol consumption, dependency, and related consequences over the past year. Each question offers 3 to 5 response options that categorize the frequency and amount of alcohol use. The total score is calculated by summing the numerical values assigned to each selected response. A total score of 8 or above indicates harmful use, while a score of 16 or above reflects a high-risk level. At the start of the study, this scale was used to include participants who scored 8 or higher. The AUDIT-C, comprising the first three items of the original AUDIT scale, was utilized as a pre-test, post-test, and follow-up assessment tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Erenköy Ruh Ve Sinir Hastaliklari Eğitim Ve Araştirma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kvamme TL, Pedersen MU, Overgaard M, Thomsen KR, Voon V. Pilot study: Improving attention bias modification of alcohol cues through concealed gaze-contingent feedback in alcohol dependence. Addict Behav Rep. 2019 Nov 6;10:100231. doi: 10.1016/j.abrep.2019.100231. eCollection 2019 Dec. PMID 31832536
- [Background] Heitmann J, van Hemel-Ruiter ME, Huisman M, Ostafin BD, Wiers RW, MacLeod C, DeFuentes-Merillas L, Fledderus M, Markus W, de Jong PJ. Effectiveness of attentional bias modification training as add-on to regular treatment in alcohol and cannabis use disorder: A multicenter randomized control trial. PLoS One. 2021 Jun 4;16(6):e0252494. doi: 10.1371/journal.pone.0252494. eCollection 2021. PMID 34086751